CLINICAL TRIAL: NCT04580186
Title: Outcome Of Classic Bladder Exstrophy Repair, Assiut University Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Eldin Anwar, assistant lecturer, Assiut University
Other Study IDs: bladder extrophy
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Bladder Exstrophy
MeSH Terms: conditions — Bladder Exstrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bladder exstrophy repair — primary complete bladder exstrophy repair

SUMMARY:
1. To review surgical and medical outcomes of the previous repaired bladder exstrophy cases.
2. To present recent developments in surgical techniques and care of these patients.

DETAILED DESCRIPTION:
* Exstrophy-epispadias complex (EEC) is a spectrum of genitourinary malformations resulting from abnormal cloacal development .
* CBE, the most common form with an incidence of 2.68 in 100,000 live births is characterized by an evaginated bladder plate, epispadias and an anterior defect of the pelvis, pelvic floor and abdominal wall
* The single most important predictor of long-term bladder growth and continence is successful primary bladder closure .
* The staged reconstruction of bladder exstrophy was proposed by Jeff and led to significant improvements in continence and renal function with excellent cosmetic results.
* The initial staged management consisted of newborn bladder and posterior urethral closure followed by bladder neck reconstruction at 2 to 3 years of age and later epispadias repair.
* The understanding that appropriately timed epispadias repair may lead to enhancement in bladder capacity led to performance of epispadias repair at 2 to 3 years of age followed by later bladder neck reconstruction. The current modification of the staged repair consists of secure bladder and posterior urethral closure in infancy followed by epispadias repair at 6 to 12 months of age and bladder neck reconstruction when the patient is able to cooperate in a good voiding program.
* Complete repair surgery is performed in a single procedure that closes the bladder and the abdomen and repairs the urethra and outer sex organs
* A failed classic bladder exstrophy (CBE) closure is defined by wound dehiscence, bladder prolapse, bladder outlet obstruction, or formation of a vesicocutaneous fistula.

ELIGIBILITY:
Inclusion Criteria:

- All patient with CBE who underwent repair at Assiut university hospital.

Exclusion Criteria:

* Cloacal exstrophy isolated epispadias previous failed repair out Assiut university hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: : patients with bladder exstrophy attending assiut university urology hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate results of the technique used for bladder exstrophy repair | base line
  complete bladder exstrophy repair

SECONDARY OUTCOMES:
Present recent development in care and repair of these patients | baseline
  update in surgical technique

REFERENCES:
- [Background] Jayachandran D, Bythell M, Platt MW, Rankin J. Register based study of bladder exstrophy-epispadias complex: prevalence, associated anomalies, prenatal diagnosis and survival. J Urol. 2011 Nov;186(5):2056-60. doi: 10.1016/j.juro.2011.07.022. Epub 2011 Sep 25. PMID 21944104
- [Background] Mayo C, Hendricks W. Exstrophy of the bladder. Surg Gynecol Obstet. 1926;43:129-34.
- [Background] Jeffs RD. Functional closure of bladder exstrophy. Birth Defects Orig Artic Ser. 1977;13(5):171-3. No abstract available. PMID 588684
- [Background] Chan DY, Jeffs RD, Gearhart JP. Determinants of continence in the bladder exstrophy population: predictors of success? Urology. 2001 Apr;57(4):774-7. doi: 10.1016/s0090-4295(00)01102-x. PMID 11306402
- [Background] Novak TE, Costello JP, Orosco R, Sponseller PD, Mack E, Gearhart JP. Failed exstrophy closure: management and outcome. J Pediatr Urol. 2010 Aug;6(4):381-4. doi: 10.1016/j.jpurol.2009.10.009. Epub 2009 Nov 10. PMID 19906564